CLINICAL TRIAL: NCT02050243
Title: The Use of 5-aminolevulinic Acid (ALA) as an Intraoperative Tumor Marker for Resection of Pediatric CNS Tumors
Brief Title: The Use of 5-aminolevulinic Acid (ALA) as an Intraoperative Tumor Marker for Resection of Pediatric Central Nervous System (CNS) Tumors
Acronym: 5-ALA
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Principal Investigator, michal roll, research and development director, Tel-Aviv Sourasky Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TASMC-13-JR-528-CTIL
Record Dates: First submitted 2013-11-20; First posted 2014-01-30 (Estimated); Last update posted 2014-01-30 (Estimated); Status verified 2014-01

CONDITIONS: Central Nervous System Tumor, Pediatric
Keywords: pediatrics; brain tumor; CNS; fluorescence; 5ALA
MeSH Terms: conditions — Central Nervous System Neoplasms; Brain Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 5ALA (Experimental): All included patients will receive 20mg/kg of 5ALA (oral suspension) about 3 hours prior to surgery
  Interventions: Drug: 5ALA

INTERVENTIONS:
Drug: 5ALA — 20mg/kg of oral suspension of 5ALA

SUMMARY:
Surgery is the cornerstone treatment of most pediatric CNS tumors, including astrocytomas, ependymomas, medulloblastomas, and many other pathologies.

In most pediatric CNS tumors, the aim of surgery is maximal tumor resection, while preserving neurological function. Extent of tumor residual has been shown to be a major prognostic factor for progression free survival (PFS), and survival in several malignant and low-grade tumors such as medulloblastomas, ependymomas, and astrocytic tumors.

5-aminolevulinic acid (5-ALA) has been shown to be valuable in intraoperative marking of various cancers. Following oral admission, during surgery, the tumor tissue is illuminated by blue light. Tumor cells tend to metabolize 5-ALA to a porphyrin named protoporhyrin IX (PpIX). PpIX reacts with the blue light and emits a pinky color (- fluorescence). This enables the surgeon to better identify tumor cells and perform a more extensive resection.

Over recent years, many studies have proven the efficacy using 5-ALA for resecting various intracranial and spinal tumors, thus achieving a better tumor control.

In the suggested study, we propose using the same technique for various pediatric central nervous system tumors.

We will focus on the correlation between various pathologies and the fluorescence, trying to deduce the role of 5-ALA in resection of specific pathologies.

Also, we will study the safety of 5-ALA use in the pediatric population.

DETAILED DESCRIPTION:
Following the above general description, eligible children will receive 5-aminolevulinic acid (5ALA) prior to surgery.

During surgery, careful attention will be payed to the fluorescence from the tumor, as well as the ability to differentiate between tumor and non tumorous tissue.

Comparisons between fluorescence and pathologies will be performed. Additionally, careful documentation of side effects will be done, to increase the safety of 5ALA use.

ELIGIBILITY:
Inclusion Criteria:

* Age 3 -18 years old
* Any CNS related pathology (including intraaxial and extraaxial tumors, intracranial or spinal intradural) that is planned for either open (microscopic) resection (or biopsy), or lesions undergoing stereotactic biopsies.
* Parental consent
* No personal or familial (1st degree) history of porphyria
* Liver function test within normal limits (alanine aminotransferase (ALT), aspartate aminotransferase (AST)<2 * upper normal limit)
* Normal renal function (Cr <2)

Exclusion Criteria:

* Surgery with no microscopic use (i.e. purely endoscopic surgeries)
* History of hepatic disease within last 12 months
* History of cutaneous photosensitivity, hypersensitivity to porphyrins, photodermatosis, exfoliative dermatitis, or porphyria
* Inability to comply with photosensitivity precautions

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2014-02; Primary Completion 2016-02 (Estimated); Study Completion 2017-02 (Estimated)

PRIMARY OUTCOMES:
sensitivity of 5ALA fluorescence to intraoperatively detect pediatric CNS tumor tissue | up to 2 weeks
  about 3hour following the 5ALA admission, the patient undergoes surgery. during surgery, global impression of tumor fluorescence will be appreciated (none, inhomogenous, intense homogenous) additionally, tumor samples will be taken from various regions, including various fluorescence regions, to try and correlate tumor regions (e.g. necrosis and viable tumor) with fluorescence (and measure the sensitivity of the 5ALA to the specific tumor)
number of patients with 5ALA related side effects | 2 weeks
  5ALA is known to cause skin hypersensitivity reaction following direct sun light exposure, during the first 48 hours after admission. also, transient elevation in liver enzymes have been documented.
  the investigators will supervise these reactions during the postoperative phase

CONTACTS AND LOCATIONS:
Locations (1):
- Department of pediatric neurosurgery, Tel Aviv, Israel, Israel